CLINICAL TRIAL: NCT03632421
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Respiratory Symptoms Substudy of ESTxENDS
Brief Title: The ESTxENDS Trial- Substudy on the Effects of Using Electronic Nicotine Delivery Systems (ENDS/Vaporizer/E-cig) on Respiratory Symptoms
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332a
Record Dates: First submitted 2018-06-25; First posted 2018-08-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Respiratory Disease
MeSH Terms: conditions — Smoking Cessation; Respiration Disorders

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Respiratory symptoms outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland. Cigarette smoking eventually kills one in two smokers, mostly through cancer, heart disease and respiratory failure. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking.

Studies suggest that ENDS use improves health outcomes, such as reducing respiratory symptoms, and presents only minimal respiratory risks, such as mild throat irritation and dry cough.

In a prospective 6-month randomized, controlled trial evaluating smoking reduction/abstinence in 300 smokers not intending to quit experimenting two different nicotine strengths of a e-cigarette model compared to its non-nicotine choice, respiratory symptoms similarly improved in all three study groups. One study compared the short-term effects of cigarette smoking to ENDS use and found that cigarette smoking led to an acute reduction in lung function, which was not observed with ENDS. Findings on short-term airway resistance is conflicting. Short term increase in resistance in ENDS users might be caused by aerosolizing the liquid, and not by the same substances that harm lung function in cigarette smokers. Smokers who shifted from tobacco cigarettes to ENDS have offered anecdotes of dramatically improved lung function, but animal models suggest that ENDS liquids can increase markers of asthma. No large randomized trials have tested the effect of ENDS on respiratory symptoms.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-months period. Respiratory symptoms such as chronic obstructive pulmonary disease (COPD), asthma and dyspnea will be assessed by means of questionnaires at baseline and at 6-, 12- and 24-months follow up. This trial will provide useful data on changes in respiratory symptoms in a large sample of participants.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Assessment of respiratory symptoms (Chronic obstructive pulmonary disease (COPD)_1 | 6 months post quit date
  Measured using COPD assessment test (CAT). The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The CAT has 8 items and the scaling of each item is from 1 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Assessment of respiratory symptoms (Chronic obstructive pulmonary disease (COPD)_2 | 12 months post quit date
  Measured using COPD assessment test (CAT). The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The CAT has 8 items and the scaling of each item is from 1 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Assessment of respiratory symptoms (Chronic obstructive pulmonary disease (COPD)_3 | 24 months post quit date
  Measured using COPD assessment test (CAT). The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The CAT has 8 items and the scaling of each item is from 1 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Assessment of respiratory symptoms (Dyspnea)_1 | 6 months post quit date
  Measured using mMRC- Dyspnea scale. The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4.
Assessment of respiratory symptoms (Dyspnea)_2 | 12 months post quit date
  Measured using mMRC- Dyspnea scale. The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4.
Assessment of respiratory symptoms (Dyspnea)_3 | 24 months post quit date
  Measured using mMRC- Dyspnea scale. The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4.
Assessment of respiratory symptoms (Asthma)_1 | 6 months post quit date
  Measured using the Asthma Control Test ACT and questions from the European community respiratory health survey ECRHS. The ACT is self-administered tool with 5-items assessing the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scaling of items is on a 5-point scale. The scores range from 5 to 25, with higher scores reflecting greater asthma control.
Assessment of respiratory symptoms (Asthma)_2 | 12 months post quit date
  Measured using the Asthma Control Test ACT and questions from the European community respiratory health survey ECRHS. The ACT is self-administered tool with 5-items assessing the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scaling of items is on a 5-point scale. The scores range from 5 to 25, with higher scores reflecting greater asthma control.
Assessment of respiratory symptoms (Asthma)_3 | 24 months post quit date
  Measured using the Asthma Control Test ACT and questions from the European community respiratory health survey ECRHS. The ACT is self-administered tool with 5-items assessing the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scaling of items is on a 5-point scale. The scores range from 5 to 25, with higher scores reflecting greater asthma control.

SECONDARY OUTCOMES:
Change in respiratory symptoms (Chronic obstructive pulmonary disease (COPD) | Change from baseline to 6,12, 24 months post quit date
  Measured using COPD assessment test (CAT). The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The CAT has 8 items and the scaling of each item is from 1 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Change in respiratory symptoms (Dyspnea) | Change from baseline to 6,12, 24 months post quit date
  Measured using mMRC- Dyspnea scale. The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4.
Change in respiratory symptoms (Asthma) | Change from baseline to 6,12, 24 months post quit date
  Measured using the Asthma Control Test ACT and questions from the European community respiratory health survey ECRHS. The ACT is self-administered tool with 5-items assessing the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scaling of items is on a 5-point scale. The scores range from 5 to 25, with higher scores reflecting greater asthma control.
Assessment of adverse respiratory effects due to ENDS use | 1 week post quit date
  Adverse respiratory effects due to ENDS use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due to ENDS use | 2 weeks post quit date
  Adverse respiratory effects due to ENDS use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due to ENDS use | 4 weeks post quit date
  Adverse respiratory effects due to ENDS use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due to ENDS use | 8 weeks post quit date
  Adverse respiratory effects due to ENDS use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due to ENDS use | 6,12, 24 months post quit date
  Adverse respiratory effects due to ENDS use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | Baseline
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | 1 week post quit date
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | 2 weeks post quit date
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | 4 weeks post quit date
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | 8 weeks post quit date
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | 6,12, 24 months post quit date
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.
Assessment of adverse respiratory effects due tobacco cigarette use | Change from baseline to 6,12, 24 months post quit date
  Adverse respiratory effects due to tobacco cigarette use use are assessed using questionnaires or over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin; Universität Bern
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Jha P, Ramasundarahettige C, Landsman V, Rostron B, Thun M, Anderson RN, McAfee T, Peto R. 21st-century hazards of smoking and benefits of cessation in the United States. N Engl J Med. 2013 Jan 24;368(4):341-50. doi: 10.1056/NEJMsa1211128. PMID 23343063
- [Background] Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. Ther Adv Drug Saf. 2014 Apr;5(2):67-86. doi: 10.1177/2042098614524430. PMID 25083263
- [Background] Caponnetto P, Campagna D, Cibella F, Morjaria JB, Caruso M, Russo C, Polosa R. EffiCiency and Safety of an eLectronic cigAreTte (ECLAT) as tobacco cigarettes substitute: a prospective 12-month randomized control design study. PLoS One. 2013 Jun 24;8(6):e66317. doi: 10.1371/journal.pone.0066317. Print 2013. PMID 23826093
- [Background] Flouris AD, Chorti MS, Poulianiti KP, Jamurtas AZ, Kostikas K, Tzatzarakis MN, Wallace Hayes A, Tsatsakis AM, Koutedakis Y. Acute impact of active and passive electronic cigarette smoking on serum cotinine and lung function. Inhal Toxicol. 2013 Feb;25(2):91-101. doi: 10.3109/08958378.2012.758197. PMID 23363041
- [Background] Vardavas CI, Anagnostopoulos N, Kougias M, Evangelopoulou V, Connolly GN, Behrakis PK. Short-term pulmonary effects of using an electronic cigarette: impact on respiratory flow resistance, impedance, and exhaled nitric oxide. Chest. 2012 Jun;141(6):1400-1406. doi: 10.1378/chest.11-2443. Epub 2011 Dec 22. PMID 22194587
- [Background] Lim HB, Kim SH. Inhallation of e-Cigarette Cartridge Solution Aggravates Allergen-induced Airway Inflammation and Hyper-responsiveness in Mice. Toxicol Res. 2014 Mar;30(1):13-8. doi: 10.5487/TR.2014.30.1.013. PMID 24795794